CLINICAL TRIAL: NCT05747651
Title: 3TR (Taxonomy, Treatment, Targets and Remission) Systemic Lupus Erythematosus Study Protocol 2
Acronym: 3TR-SLE2
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC22.1068 (3TR-SLE2)
Record Dates: First submitted 2023-01-30; First posted 2023-02-28 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic; Lupus; Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Active SLE: Patients will undergo regular follow-up where routine clinical examination and laboratory assessments will be conducted, and biological samples will be obtained. The patients will be instructed to contact their center whenever they develop a symptom suspicious of flare. In such cases, an unscheduled visit will be conducted for clinical examination, assessment and sampling similar to the last visit.
  If a patient needs a major change in therapy at one of the scheduled visits or at an unscheduled visit, an early termination (ET) visit will be planned. Patients requiring a major change in therapy due to active disease (defined as BILAG A or B) from week 12 through week 52 will undergo two additional evaluations at week +26 and at week +52 from the time of early termination/new therapy initiation in order to determine biomarkers of secondary response after the change in therapy (herein termed secondary response) and persistent non- response (herein termed refractory disease).
  Interventions: Biological: Blood sample; Biological: Urine sample; Biological: Saliva sample; Biological: Stool sample; Biological: Tissue sample

INTERVENTIONS:
Biological: Blood sample — Total volume of blood (on each sampling occasion): 54,5mL.
Biological: Urine sample — Urine: 100 mL which will be centrifuged. The pellet will be frozen, and the urine supernatant will be aliquoted.
Biological: Saliva sample — Saliva: will be collected in special container for saliva microbiome and methylation.
Biological: Stool sample — Stool: One sample for microbiome to be sent to the biobank, frozen at -80 °C.
Biological: Tissue sample — Tissue samples for organ-specific manifestations:
  * Kidney tissue in lupus nephritis: one small fragment of the fresh kidney biopsy will be stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.
  * Skin tissue (at selected centers) from inflamed lesion and non-inflamed skin from the gluteal region will be obtained through punch biopsy and stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.
  * Synovial tissue (at selected centers) will be obtained through ultrasound-directed arthroscopy and stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.
  * Aspirate from swollen lymph nodes (at selected centers) will be obtained and stored in a 10% dimethyl sulfoxide (DMSO) solution (slow freezing to -80 °C) until shipment.

SUMMARY:
The natural history of Systemic lupus erythematosus (SLE) is characterized by relapses or flares alternated with periods of remission. Flares are associated with accrual of organ damage independently of other risk factors, both contributing to a considerable morbidity. No useful biomarker is currently available to predict which patients with a quiescent disease are at risk of flare.

The 3TR project (funded by the Innovative Medicines Initiative 2 Joint Undertaking under grant agreement No 831434, and supported by European Union's Horizon 2020 research and innovation programme and EFPIA) is a transdisciplinary consortium that primary aims at identifying biosignatures as predictors of response and non-response to therapy in seven different autoimmune, allergic and inflammatory diseases, including SLE. 3TR will perform a longitudinal multi-dimensional molecular analysis in patients with these diseases. A molecular profiling approach is a modern and innovative way to investigate and stratify heterogeneous diseases on the basis of their common biomolecular pathways. The main hypothesis of the 3TR project is that data obtained from multiomic analysis across the seven different diseases will identify shared biological pathways that better predict the response or non-response to therapy despite their differences in terms of clinical phenotypes and pathogenetic mechanisms. Therefore patients from multiple European centers participating in 3TR will be recruited for a longitudinal clinical follow-up and collections of several samples that will be used to perform multi-omic analysis.

DETAILED DESCRIPTION:
The study will be carried out in the framework of the IMI2 (innovative medicine initiative) and EFPIA (European Federation of Pharmaceutical Industries and Associations)-funded 3TR (Taxonomy, Treatment, Targets and Remission) project. The programme is supported by the European Union's Horizon 2020 research and innovation programme. 3TR is funded under the grant agreement No 831434 and it runs from 2019 to 2026.

3TR is a transdisciplinary consortium that aims to perform a longitudinal multi-dimensional molecular analysis in patients with autoimmune, allergic and inflammatory diseases. A molecular profiling approach is a modern and innovative way to investigate and stratify heterogeneous diseases on the basis of their common biomolecular pathways. The main hypothesis of the 3TR project is that data obtained from multiomic analysis across seven different diseases, including SLE, will identify shared biological pathways that better predict the response or non-response to therapy despite their differences in terms of clinical phenotypes and pathogenetic mechanisms. Patients from multiple European centers participating in 3TR will be recruited for a longitudinal clinical follow-up and collections of several samples that will be used to perform multi-omic analysis.

Several innovations are expected within the 3TR project to increase the knowledge of pathogenetic mechanisms underlying the clinical phenotypes in SLE, and to unravel, in the complexity of SLE biomolecular heterogeneity, the pathways of response or non-response to treatment, as well as, at an earlier stage, the processes that may lead to disease flare. These insights could ultimately allow the possibility to effectively practice prevention and counselling, to adopt measures of personalized treatment or to perform drug repurposing using the knowledge gained from the SLE studies and the studies on other diseases within the 3TR project.

Moreover, the impact of the COVID-19 viral pandemic will be implemented in the research. More specifically, the investigators will study the impact of the presence of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on the development of flare, as well as on the response or non-response to immunomodulatory therapy.

To implement the strategy, a two-step research has been designed, and comprises: 1. The flare biomarker study (3TR SLE 1) is considered a "feeding" phase before the main part. Patients who meet the inclusion criteria for 3TR SLE 2 will be proposed to participate in the second study. 2. The response biomarker study (3TR SLE 2), which is a prospective study (main part). The present protocol relates to the response biomarker study (3TR SLE 2).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age at the time of inclusion ≥ 18 years.
* 2. Able to consent and agree to participate in the study.
* 3. Diagnosis of SLE according to the EULAR/ACR criteria.
* 4. Patients should have at least one of the following: i. active arthritis, attributed to SLE (BILAG A or B in the musculoskeletal domain).

ii. active skin disease, attributed to SLE (BILAG A or B in the mucocutaneous domain).

iii. active biopsy-proven lupus nephritis (LN; ISN/RPS class III, IV or V), with or without extrarenal organ involvement.

iv. active CNS involvement as a main manifestation (with or without other organ involvement) along with initiation of new treatment for CNS involvement (BILAG A or B in the neuropsychiatric domain).

* 5. Stable standard therapy for at least 30 days, including hydroxychloroquine (HCQ) or chloroquine treatment, unless contraindicated or documented intolerance.

Exclusion Criteria:

* 1. Serological activity only without signs of clinically active disease.
* 2. Pregnancy and/or breastfeeding.
* 3. Unable/unaware to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SLE patients with active disease, defined as a BILAG A or B within certain domains (see inclusion criteria) will be included in this study. These patients will either be directly recruited to this study or originate from the "feeding" phase (3TR-SLE, flare biomarker study, NCT05458622) when a flare is detected. There will be no restriction regarding current or previous therapies.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) response at week 52 from baseline, including SLEDAI-2K, CLASI-A, OCS dosage reduction, and patient-reported outcomes. | 52 weeks

SECONDARY OUTCOMES:
SLE Responder Index (SRI)-4, SRI-5 and SRI-6 response (at all time points) | 52 weeks
  The outcome measure correponds to an improve of at least 4, 5 or 6 of SLEDAI-2K score, no aggravation of BILAG A or B score and no aggravation of the PhGA.
Time to BICLA response. | 52 weeks
Time to SRI response. | 52 weeks
Failure to attain BICLA response (at all time points). | 52 weeks
  The BICLA measurement has no unit.
Failure to attain SRI-4, SRI-5 and SRI-6 response (at all time points). | 52 weeks
  The outcome measure correponds to a failure to attain at least 4, 5 or 6 of SLEDAI-2K score, no aggravation of BILAG A or B score and no aggravation of the PhGA.
Change in SLEDAI-2K scores (at all time points). | 52 weeks
  The change in the SLEDAI-2K is a number without unit to see change in the SLEDAI score. The SLEDAI score is obtained on a scale 0-115.
Change in Physician's Global Assessment (PhGA, on a scale 0-3) (at all time points). | 52 weeks
  The Physician's Global Assessment (PhGA) is a number without unit on a scale 0-3.
Change in Patient's Global Assessment (PGA, on a 0-10 VAS) (at all time points). | 52 weeks
  The Patient's Global Assessment (PGA) is a patient assessment without unit on a scale 0-10.
Lupus Low Disease Activity State (LLDAS), and its individual components (at all time points). | 52 weeks
  The Lupus Low Disease Activity State (LLDAS) is assessed as "present" or "absent".
Remission according to DORIS, and its individual components (at all time points). | 52 weeks
  The Remission according to DORIS is assessed as "present" or "absent". DORIS is a score obtained when patient has 0mg of corticoisteroids and a stable treatment with no activity of the disease.
Flare, based on BILAG (any new worsening in BILAG, or any new BILAG A or B) or SELENASLEDAI Flare Index (SFI) (at all time points). | 52 weeks
  The flare based on BILAG is assessed as "yes" or "no".
Renal response/non-response, according to the 2019 EULAR/EDTA recommendations. | 52 weeks
Organ-specific outcome measures with CLASI for mucocutaneous involvement (at all time points). | 52 weeks
  The CLASI activity is ranged from 0-70, with higher scores indicating more severe skin disease. It evaluates through 13 anatomical regions erythema and scale hypertrophy (from 0 to 3 and 0 to 2 respectively). The activity scores of 0-9 indicating mild disease, 10-20 indicating moderate disease, and 21-70 indicating severe disease. It is also a useful tool in determining whether or not patients responded to treatment, as patients who improved clinically had a mean a 4-point or 20% decrease in the CLASI activity score to identify improvement.
Organ-specific outcome measures with 44 joint assessment of tender and swollen joints for articular involvement (at all time points). | 52 weeks
Worsening in SLICC/ACR Damage Index (SDI) score (at week 52). | 52 weeks
  The Worsening in SLICC/ACR Damage Index (SDI) score is assessed by a binary response as "present" or "absent". The SLICC/ACR Damage Index (SDI) is the score of the damage of the disease and is a number out of 46 without unit.
Health-related quality of life (HRQoL) assessed with EQ-5D-5L (at week 26 and week 52). | 52 weeks
  EQ-5D-5L evaluates health-related quality of life via a descriptive system and a visual analogue scale. The descriptive system comprises a list of quotes divided in five dimensions: mobility, self-care, usual activities, pain and discomfort and anxiety and depression. For each dimension, the patient choses a level of severity of his/her condition by selecting one quote among five propositions. The visual analogue scale is used for the patient to rate his/her general health condition on a scale of 1 to 100.
Health-related quality of life (HRQoL) assessed with FACIT-F (at week 26 and week 52). | 52 weeks
  FACIT-F is a tool to assess tiredness where the patient tiredness is rated by replying to 13 quotes on a 5-point scale going from "not at all" to "very much".
Health-related quality of life (HRQoL) assessed with Medical Outcomes Study 36-item Short Form health survey (SF-36) (at week 26 and week 52). | 52 weeks
  SF-36 is a patient-reported short form health survey composed of 36 items.
Health-related quality of life (HRQoL) assessed with Epworth Sleepiness scale (ESS) (at week 26 and week 52). | 52 weeks
  The ESS is a self-administered questionnaire with 8 questions where patients are asked to rate on a 4-point scale (0-3) their usual chances of dozing off or falling asleep while engaged in eight different activities.
Health-related quality of life (HRQoL) assessed with Lupus-QoL (at week 26 and week 52). | 52 weeks
  The LupusQoL is a lupus-specific HRQOL questionnaire consisting of 34 items grouped in eight domains: physical health, pain, planning, intimate relationships, burden to others, emotional health, body image and fatigue. A score from 0 to 100 (best HRQOL) is calculated for each domain.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of or time to BICLA. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of or time to the British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA). BICLA is a validated composite global measure of SLE disease activity including SLEDAI-2K, CLASI-A, OCS dosage reduction, and patient-reported outcomes.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of or time to SLE Responder Index (SRI). | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of or time to SRI. SRI is an index to evaluate the activity of the disease.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of LLDAS. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of Lupus Low Disease Activity State (LLDAS). Low disease activity is obtained when patient has 7.5 mg of corticosteroids and stable immunosuppressive treatement ans stability of the disease.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of DORIS. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of DORIS. DORIS is a score obtained when patient has 0 mg of corticoisteroids and a stable treatment with no activity of the disease. DORIS is assessed as "present" or "absent".
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of SLEDAI-2K. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of SLEDAI-2K. SLEDAI-2K is a number without unit on a 0 to 105-scale.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of PhGA. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment PhGA. The Physician's Global Assessment (PhGA) is a number without unit.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of PGA. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of PGA. The Patient's Global Assessment (PGA) is a number without unit.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on SDI scores. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on SDI score. SDI score is the score of the damage of the disease and is a number out of 46 without unit.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on attainment of change in organ specific index scores. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on organ specific index scores. The organ specific index scores are scores without unit.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on Health-related quality of life (HRQoL) assessed with EQ-5D-5L. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on HRQoL assessed with EQ-5D-5L. EQ-5D-5L evaluates health-related quality of life via a descriptive system and a visual analogue scale. The descriptive system comprises a list of quotes divided in five dimensions: mobility, self-care, usual activities, pain and discomfort and anxiety and depression. For each dimension, the patient choses a level of severity of his/her condition by selecting one quote among five propositions. The visual analogue scale is used for the patient to rate his/her general health condition on a scale of 1 to 100.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on Health-related quality of life (HRQoL) assessed with FACIT-F. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on HRQoL assessed with FACIT-F. FACIT-F is a tool to assess tiredness where the patient tiredness is rated by replying to 13 quotes on a 5-point scale going from "not at all" to "very much".
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on Health-related quality of life (HRQoL) assessed with Medical Outcomes Study 36-item Short Form health survey (SF-36). | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on HRQoL assessed with Medical Outcomes Study 36-item Short Form health survey (SF-36). SF-36 is a patient-reported short form health survey composed of 36 items.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on Health-related quality of life (HRQoL) assessed with Epworth Sleepiness scale (ESS). | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on HRQoL with Epworth Sleepiness scale (ESS). The ESS is a self-administered questionnaire with 8 questions where patients are asked to rate on a 4-point scale (0-3) their usual chances of dozing off or falling asleep while engaged in eight different activities.
Impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on Health-related quality of life (HRQoL) assessed with Lupus-QoL. | 52 weeks
  This exploratory study will observe the impact of anti-SARS-CoV-2 antibodies of different isotypes (IgA, IgG, IgM) on HRQoL assessed with Lupus-QoL. The LupusQoL is a lupus-specific HRQOL questionnaire consisting of 34 items grouped in eight domains: physical health, pain, planning, intimate relationships, burden to others, emotional health, body image and fatigue. A score from 0 to 100 (best HRQOL) is calculated for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Jousse-Joulin, Principal Investigator — CHU Brest
Locations (1):
- CHU Brest, Brest, France, France

IPD SHARING:
Plan to Share IPD: Undecided